CLINICAL TRIAL: NCT04346914
Title: Phase Ib Study of Recombinant Anti-PD-L1 Monoclonal Antibody Injection (ZKAB001) Combined With Carboplatin and Etoposide in the Treatment of Extensive Small Cell Lung Cancer
Brief Title: Study of ZKAB001 Combined With Carboplatin and Etoposide in the Extensive Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTL-LEES-2019-03
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Extensive Stage Small Cell Lung Cancer
Keywords: ES-SCLC
MeSH Terms: interventions — Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined treatment group (Experimental): recombinant anti-PD-L1 monoclonal antibody injection combined with carboplatin and etoposide ZKAB001 ,5 mg/kg, d1，q3w； carboplatin，5 AUC，d1，q3w； etoposide，100mg/m2，d1~3，q3w
  Interventions: Biological: recombinant anti-PD-L1 monoclonal antibody injection combined with carboplatin and etoposide

INTERVENTIONS:
Biological: recombinant anti-PD-L1 monoclonal antibody injection combined with carboplatin and etoposide — ZKAB001 ,5 mg/kg, d1，q3w； carboplatin，5 AUC，d1，q3w； etoposide，100mg/m2，d1~3，q3w

SUMMARY:
To evaluate the safety and efficacy of recombinant anti-PD-L1 monoclonal antibody injection (ZKAB001) combined with carboplatin and etoposide in the treatment of extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
To evaluate the safety and preliminary efficacy of recombinant anti-PD-L1（Programmed cell death ligand 1）monoclonal antibody injection (ZKAB001) combined with carboplatin and etoposide in the treatment of extensive-stage small cell lung cancer. The study will last until the number of patients who permanently stop taking drugs due to toxicity in the first two cycles is less than 1/3 of the total number of patients.

ELIGIBILITY:
Inclusion Criteria:

* both men and women, age ≥ 18 years old and ≤ 75 years old.
* histologically confirmed SCLC
* extensive stage SCLC (ES-SCLC) according to (VALG) staging of American Veterans Lung Cancer Association.
* have not received first-line systemic therapy for ES-SCLC in the past.
* surgery and adjuvant therapy for cure, such as radiotherapy and chemotherapy, were performed in the past, and there was no treatment interval of at least 6 months from the last chemotherapy, radiotherapy or radiotherapy or chemotherapy to the diagnosis of ES-SCLC.
* PS 0 or 1.
* estimated survival time > 12 weeks.
* CT or MRI scan with at least one measurable lesion less than 28 days before the first dose of the study drug (RECIST v1.1).
* male subjects and women of childbearing age must have contraception within 6 months from the beginning of the first drug study to the last study drug.
* before the first dose of the drug, the laboratory test values met the following conditions: (1) Blood routine test: WBC ≥ 3.0x10^9 / L, ANC ≥ 1.5x10^9 /L, PLT ≥ 100x10^9 /L, hGB ≥ 90g / L; (2) liver function: AST ≤ 2.5 ULN, ALT ≤ 2.5 ULN; ALT and AST < 5 ULN for liver metastases; TBIL ≤ 1.5 ULN; ALB ≥ 30 g L; (3) Renal function: serum creatinine ≤ 1.5 ULN or creatinine clearance rate (Ccr) ≥ 40 mL/min (Cockcroft/Gault formula); (4) Coagulation function: INR ≤ 1.5, APTT ≤ 1.5 ULN; (5) ALP ≤ 2.5 ULN, ALP ≤ 5 ULN. for bone metastasis subjects,
* tumor tissue samples that can meet the detection of PD-L1 expression can be provided during the screening period and within 4 weeks after selection.
* voluntarily sign informed consent form (ICF)

Exclusion Criteria:

* before entering the group, the patients received any T cell co-stimulatory or immune checkpoint inhibitors, including, but not limited to, cytotoxic T lymphocyte associated antigen-4 (CTLA-4) inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors or other drugs targeting T cells; previously received anti-vascular endothelial growth factor (VEGF) or vascular endothelial growth factor receptor (VEGFR) therapy.
* active brain metastasis or meningeal metastasis.
* Patients with brain metastasis after treatment need to meet the following conditions: asymptomatic; no imaging evidence of progress ≥ 4 weeks after treatment; completion of treatment within 14 days before the first dose of the study drug; and no need to receive systemic corticosteroids (> 10mg/ prednisone or equivalent) less than 14 days before the first dose of the study drug.
* radiotherapy for the chest and whole brain was completed less than 4 weeks before the first dose of the study drug (palliative radiotherapy for bone lesions is allowed ).
* the third space effusion with clinical symptoms, such as pericardial effusion, pleural effusion and peritoneal effusion which cannot be controlled by pumping or other treatment.
* active, known or suspected autoimmune diseases. Patients with vitiligo, type I diabetes, residual hypothyroidism caused by autoimmune thyroiditis that only require hormone replacement therapy, or are not expected to recur in the absence of external stimulation can be included in the group.
* corticosteroids (> 10 mg/ prednisone or equivalent dose) or other immunosuppressants were used within 14 days before the first study.

Inhalation or topical use of steroids and adrenal replacement steroids are allowed in the absence of active autoimmune disease; for patients receiving short-term, systemic immunosuppressive therapy, for example, glucocorticoids for nausea, vomiting, or allergic reaction management or preventive use can be admitted after consultation with the sponsor. Allow the use of salt corticosteroids in the treatment of postural hypotension and the use of low-dose glucocorticoid supplements in the treatment of adrenocortical insufficiency;

* subjects who had been vaccinated or planned to receive live vaccines within 4 weeks before the first study.
* Interstitial pneumonia (ILD) disease, drug-induced pneumonia, radiation pneumonia requiring steroid treatment or active pneumonia with clinical symptoms.
* active pulmonary tuberculosis or screening subjects with a history of active pulmonary tuberculosis infection within 1 year before treatment, whether treated or not.
* except for alopecia and fatigue, other toxicities caused by previous antineoplastic therapy need to be restored to CTCAE 5.0 ≤ 1 before the first dose. Some other toxicities caused by previous antineoplastic therapy are not expected to be resolved and have long-term persistent sequelae, such as neurotoxicity caused by platinum-based therapy, which are allowed to be included in the group.
* uncontrolled hypertension (systolic blood pressure ≥ 140mmHg and / or diastolic blood pressure ≥ 90 mmHg), history of hypertensive crisis or hypertensive encephalopathy.
* there are uncontrolled clinical symptoms or diseases of the heart, such as: (1)heart failure defined by New York Heart Association (NYHA)in grade 2 or above (2) unstable angina pectoris (3) myocardial infarction within 6 months (4) clinically significant supraventricular or ventricular arrhythmias need to be treated.
* uncontrolled active infections (e.g. need intravenous antibiotics, antifungal or antiviral therapy).
* HIV infection, HBsAg positive and peripheral blood HBV-DNA titer ≥ 0.5 × 10^3 copies / mL or HCV positive (HCV RNA or HCV Ab test indicated acute or chronic infection).
* pregnant or lactating women.
* known allergies to study drugs or excipients, and known severe allergic reactions to any monoclonal antibody; allergic history of carboplatin or etoposide.
* other malignant tumors occurred less than 5 years before the first dose, except for fully treatable cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection, ductal carcinoma in situ after radical resection, and breast cancer without recurrence and metastasis after radical resection.
* known cases of mental illness, alcohol abuse, inability to quit smoking, drug use or substance abuse.
* have been treated with any other experimental drugs or participated in another interventional clinical study within 4 weeks before signing ICF

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-08 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
DLT | 28 days after first dose
  The number of patients who permanently stop taking drugs due to toxicity is less than 1/3 of the total number of patients.

SECONDARY OUTCOMES:
objective response rate | 12 months
  Percentage of patients in partial and complete response
progression free survival | 12 months
  time between first dose of study drug to disease progression
The positive rate of PD-L1 expression in tumor tissue | 12 months
  The positive rate of PD-L1 expression in tumor tissue.
The positive rate of anti-drug antibody (ADA); | 12 months
  The positive rate of anti-drug antibody (ADA);
overall survival | 12 months
  time between first dose of study drug to death caused by any reason

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu S, Chen Z, Cui J, Guo R, Li Z, Li BX, Dai X. Efficacy and Safety of Anti-Programmed Death-Ligand 1 Monoclonal Antibody Socazolimab With Carboplatin and Etoposide for Extensive-Stage SCLC: Results From the Phase 1b Clinical Trial. JTO Clin Res Rep. 2023 Feb 28;4(4):100478. doi: 10.1016/j.jtocrr.2023.100478. eCollection 2023 Apr. PMID 37020926